CLINICAL TRIAL: NCT03954899
Title: Evaluating the Disease Modifying Potential of a Sleep Intervention on Alzheimer's Disease (AD) Biomarkers
Brief Title: Disease Modifying Potential of 5mg of Melatonin on Cognition and Brain Health in Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natalie Denburg (Other)
Responsible Party: Sponsor-Investigator, Natalie Denburg, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201903824; 1R01AG062673-01 (NIH)
Record Dates: First submitted 2019-05-15; First posted 2019-05-17 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Mild Cognitive Impairment; Cognitive Decline; Healthy Aging
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- MCI+ Melatonin 5mg (Experimental): MCI+ individuals receiving 5mg of melatonin-OTC for a period of 9 months
  Interventions: Dietary Supplement: melatonin
- MCI+ placebo (Placebo Comparator): MCI+ individuals receiving placebo for a period of 9 months
  Interventions: Other: placebo
- MCI- Melatonin 5mg (Experimental): MCI- individuals receiving 5mg of melatonin-OTC for a period of 9 months
  Interventions: Dietary Supplement: melatonin
- MCI- placebo (Placebo Comparator): MCI- individuals receiving placebo for a period of 9 months
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: melatonin — 5mg of melatonin-otc 30 minutes before sleep
  Arms: MCI+ Melatonin 5mg; MCI- Melatonin 5mg
Other: placebo — placebo 30 minutes before sleep
  Arms: MCI+ placebo; MCI- placebo

SUMMARY:
The study will examine whether 5mg melatonin (over the counter, OTC) over a 9-month period improves Alzheimer's disease (AD) biomarkers and cognitive function in two groups of individuals: those with mild cognitive impairment (MCI+) and those who are not (MCI-). AD biomarkers will be measured from cerebrospinal fluid (CSF) obtained from lumbar punctures. Cognitive function will be evaluated with routine neuropsychological tests.

AS OF AUGUST 2024, THE LUMBAR PUNCTURE PROCEDURES FOR THIS CLINICAL TRIAL HAVE BEEN ELIMINATED. THAT IS, PARTICIPANTS ARE NO LONGER RECEIVING A LUMBER PUNCTURE. BUT ARE CONTINUING TO RECEIVE TWO SEPARATE BLOOD DRAWS FOR BIOMARKER TESTING.

DETAILED DESCRIPTION:
To address these broad aims, participants will be recruited from the Neuropsychology Clinic, community, Alzheimer's association local chapter events and support groups, senior citizen centers. Following fulfillment of several inclusionary and exclusionary criteria online/on the phone, participants will first complete a baseline visit with several tests designed to measure aspects of motor, affective, and cognitive function. The baseline visit will be briefer for those who do not fulfill in-person components of the inclusionary/exclusionary criteria (BMI<35; MoCA>=18; and CDR <=.5).

Based on the information obtained during the baseline visit, participants' cognitive status will be categorized as either MCI+ or MCI-. The criteria adopted in this study for a determination of MCI is less stringent than typical clinical criteria. This information will be used to conduct stratified randomization of participants to placebo or active (5mg melatonin) arms. The schedule of randomization will be determined by University of Iowa Hospital & Clinic's pharmacy so that study personnel and participants will not know which participant has been assigned to which study arm.

At the end of the baseline visit, participants will be given actigraphy watches to wear for a period of 8 weeks, a wash-out phase; phase#1. The watches monitor sleep and circadian rhythm in each participant's daily life. At the end of 8 weeks, participants will return to the lab to complete a brief battery of cognitive tests. At the end of the visit, they will be given freshly charged actigraphy watches to take home with them until week-16 as well as the first supply of study issued medications (beginning phase#2 of the study). They will receive a phone call at the beginning of week-9 to complete brief questionnaires regarding sleep quality, mood, and any physical symptoms that may be associated with study-issued medications. At the week-16 visit, the participants will return their actigraphy watches, complete brief cognitive testing, questionnaires on sleep quality, mood, physical symptoms that may be associated with study-issued medications, and complete the first LP and blood draw. They will also be given their supply of study-issued medications for the next 7-month period. They will receive a phone call around week-30 (midway between week-16 and the final study visit of week-44) to inquire about sleep quality, any physical symptoms that may be associated with study-issued medications, and mood. The final study visit will take place on week-44. The visit will be very similar to the baseline visit and will include comprehensive cognitive testing, questionnaires, and an LP. Participants will also receive a phone call the day after each LP to query them about any discomfort they may be experiencing and the adequacy of over-the-counter pain medications in addressing it.

In addition to these procedures, participants will be asked to consent to banking of CSF for assaying of future biomarkers during the two study LPs.

AS OF AUGUST 2024, THE LUMBAR PUNCTURE PROCEDURES FOR THIS CLINICAL TRIAL HAVE BEEN ELIMINATED. THAT IS, PARTICIPANTS ARE NO LONGER RECEIVING A LUMBER PUNCTURE. BUT ARE CONTINUING TO RECEIVE TWO SEPARATE BLOOD DRAWS AT WEEKS 8 AND 44 FOR BIOMARKER TESTING.

ELIGIBILITY:
Inclusion Criteria:

1. between ages of 56-85 years
2. all participants must score 18 or above on Montreal Cognitive Assessment (MoCA);
3. all participants must have a clinical dementia rating (CDR) Sum of boxes <1;
4. need to be willing to undergo CSF LP on two occasions over the course of their participation,
5. need to be able and willing to stop using any prescription or non-prescription sleep aids (e.g.(e.g. Ambien, Sonata, Lunesta, Belsomra, Rozerem, Halcion, Intermezzo, Doxepin, Melatonin, etc.) for the duration of the study except for study-issued medications
6. BMI < 35 at the time of enrollment
7. willing to bring a study partner (spouse, child or friend) who knows them well to each of the four visits

AS OF AUGUST 2024, THE LUMBAR PUNCTURE PROCEDURES FOR THIS CLINICAL TRIAL HAVE BEEN ELIMINATED. THAT IS, PARTICIPANTS ARE NO LONGER RECEIVING A LUMBER PUNCTURE. BUT ARE CONTINUING TO RECEIVE TWO SEPARATE BLOOD DRAWS FOR BIOMARKER TESTING.

The exclusion criteria are:

1. Individuals with any of the following conditions/ diseases will be excluded:

   Obstructive sleep apnea (OSA) without CPAP use, chronic obstructive pulmonary disease, emphysema, major psychiatric disease (bipolar, schizophrenia), history of alcohol/drug abuse, neurodegenerative disease diagnosis (e.g. Parkinson's, Lewy body, ALS, MS), prior history of stroke or traumatic brain injury, have undergone chemotherapy in the past 2 years, have been hospitalized for injury/surgery in the past three-months.
2. CDR>=1, clinically significant depression/anxiety (GDS>=9; GAI>=9 ),
3. Participants who are on any of the following medications will be excluded: Fluvoxamine (Luvox)/ Fluoxetine (Prozac), Nifedipine (a blood pressure medication), all anti-coagulants (e.g. Warfarin, Coumadin, Heparin, , Lovenox, Xarelto, Pradaxa, etc.), anti-seizure drugs (e.g. Acetazolamide, Carbamazepine, Clobazam, Clonazepam, Gabapentin, etc.), muscle relaxants (e.g.Baclofen, Valium/ diazepam, Flexeril, etc.), or narcotic pain relievers (e.g.Codeine, Tramadol, Hydrocodone, Demerol, etc).

Ages: 56 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Episodic memory | Assessed at pre-treatment (week-8), and two post-treatment occasions: week-16 and week-44.
  Composite episodic memory performance scores will be computed based on the following tests: Auditory Verbal Learning Test (AVLT), Free & Cued Selective Reminding Test (FCSRT), Repeatable Battery for the Assessment of Neuropsychological Status (Story memory) at the week-8, week-16, and week-44 visits. Alternate forms will be used to assess performance in each of these tests across these visits to minimize practice effects. Composite scores at week-16 and week-44 visits will reference the pretreatment group mean and standard deviations to permit the detection of deviation from pre-treatment levels.

SECONDARY OUTCOMES:
Overall cognitive function | Assessed at pre-treatment (week-8), and two post-treatment occasions: week-16 and week-44.
  Composite performance scores will be computed based on the following cognitive tests: AVLT, FCSRT, RBANS-Story, Benton Visual Retention Test (BVRT), Trail Making Test (PartsA&B), and Controlled Oral Word Association (COWA) at the week-8, week-16, and week-44 visits. Alternate forms will be used to assess performance in each of these tests, when available, across these visits to minimize practice effects. Composite scores at week-16 and week-44 visits will reference the pretreatment group mean and standard deviations to permit the detection of deviation from pre-treatment levels.
p-tau/Aβ42 ratio | Assessed at pre-treatment (week-8) and one post-treatment occasion (week-44)
  Cerebrospinal values from lumbar puncture
t-tau | Assessed at pre-treatment (week-8) and one post-treatment occasion (week-44)
  Cerebrospinal values from lumbar puncture
Sleep Efficiency | Daily from actigraphy in the pre-treatment phase which lasts 8 weeks (phase#1) and daily from actigraphy in the post-treatment phase from week-9 to week-16 (phase#2).
  Daily Sleep efficiency values obtained from actigraphy during the wash-out period (weeks 1 to 8) and sleep efficiency values obtained from actigraphy during week-8 to week-16 when participants are on placebo or the active arm.
Amplitude (Mesor) of rest-activity rhythm | Daily from actigraphy in the pre-treatment phase which lasts 8 weeks (phase#1) and daily from actigraphy in the post-treatment phase from week-9 to week-16 (phase#2).
  The 30-second activity counts from actigraphy watches will be submitted to cosinor curve analyses to permit the extraction of peak amplitude per day in both phases of the study (wash-out pre-treatment from week-1 to week-8 and week-9 to week-16 post treatment, phase#2). These amplitude values will be averaged to characterize typical amplitude for each participant within each study phase.
Acrophase of rest-activity rhythm | Daily from actigraphy in the pre-treatment phase which lasts 8 weeks (phase#1) and daily from actigraphy in the post-treatment phase from week-9 to week-16 (phase#2).
  The 30-second activity counts from actigraphy watches will be submitted to cosinor curve analyses to permit the extraction of the time of day at peak amplitude per day in both phases of the study (wash-out pre-treatment from week-1 to week-8 and week-9 to week-16 post treatment, phase#2). These acrophase values will be averaged to characterize typical timing of peak amplitude for each participant within each study phase.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Denburg, Ph.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No